CLINICAL TRIAL: NCT03233880
Title: Impact of Antichlamydial Treatment on the Rate of Preeclampsia Among Egyptian Primigravidae: a Randomized Controlled Trial
Brief Title: Impact of Antichlamydial Treatment on the Rate of Preeclampsia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, ADEL SHAFIK SALAH EL-DIN, Assistant professor, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Anti Chlamydial treatment
Record Dates: First submitted 2017-07-23; First posted 2017-07-31 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Pre-Eclampsia
Keywords: chlamydia; prevention
MeSH Terms: conditions — Pre-Eclampsia; Chlamydia Infections

STUDY DESIGN:
Intervention Model Description: randomized, double blinded controlled trial
Who Masked: Participant, Care Provider
Masking Description: double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Azithromycin group (Active Comparator): Azithromycin 1Gm orally, single dose (Xithrone 500 mg two tablets, Amoun, Inc, Cairo, Egypt) will be given to pregnant women at 16/20 weeks of pregnancy
  Interventions: Drug: Azithromycin 1gm
- placebo group (Placebo Comparator): - Matching placebo orally, single dose
  Interventions: Other: PLACEBO

INTERVENTIONS:
Drug: Azithromycin 1gm — Azithromicin 1 gm oral single dose
  Other Names: anti chlamydial treatment
  Arms: Azithromycin group
Other: PLACEBO — placebo
  Arms: placebo group

SUMMARY:
This randomized, double blinded controlled trial included 1200 healthy primigravidae who attended an outpatient clinic at 16-20weeks of pregnancy. All women were randomly divided equally into two groups, group A(600 women) who received antichlamydial treatment in the form of azithromycin 1 gram single oral dose before 20 weeks of pregnancy and group B (600 women) who received no treatment(placebo). All participants were followed up for up to 6 weeks postpartum and observed for the development of preeclampsia.

DETAILED DESCRIPTION:
Preeclampsia complicates approximately 5-8% of all pregnancies and is a major cause of maternal morbidity and mortality worldwide.Its progress differs among patients; most cases are diagnosed pre-term. Preeclampsia may also occur up to six weeks post-partum. The present study included 1200 primigravidae who attended the outpatient clinic of Ain Shams University maternity Hospital in Cairo, Egypt, for routine antenatal care between July 2016 and September 2017. The study was approved by the Ethics Committee of Ain Shams University Maternity Hospital in accordance with local research governance requirements. All participating women signed an informed consent form inclusion criteria were a primigravida, singleton pregnancy, maternal age 18-35 years, and pregnancy duration 16-20 weeks at the time of study inclusion. Exclusion criteria were Women with multi-fetal pregnancy, diabetes mellitus, chronic hypertension, or chronic renal disease.Computer based Randomization codes were placed in sequentially numbered, opaque, sealed envelopes by an observer, to be opened at time of enrollment by a pharmacist in Ain Shams University Hospital who prepared the study drug and had no further involvement with the patient's care. All data were analyzed before it was determined which group was received azithromycin and which was received placebo.

* Azithromycin 1Gm orally, single dose (Xithrone 500 mg two tablets, Amoun, Inc, Cairo, Egypt) Group (A) OR
* Matching placebo orally, single dose Group (B). Preeclampsia was defined in the terms of hypertension and proteinuria. The International Society for the Study of Hypertension (ISSH) defined preeclampsia as new hypertension and new proteinuria developing after 20 weeks of gestation and regressing remotely after delivery. Hypertension is defined as diastolic arterial blood pressure ≥90 mmHg on two or more consecutive occasions, at least 4 hours apart. Proteinuria is defined as ≥ +1 on dipstick test on 2 midstream urine collections more than 4 hours apart or 24-hour urinary protein ≥ 300mg. Severe preeclampsia was defined as follows: blood pressure >160/110 mmHg on two occasions at least 6 hours apart, proteinuria >5 gm/24 hours, oliguria < 500 ml/24 hours, thrombocytopenia < 100.000/ml, cerebral visual disturbances, epigastric pain, nausea and vomiting, impaired liver function of unclear etiology or the occurrence of complications as pulmonary edema, accidental hemorrhage or fetal compromise.

ELIGIBILITY:
Inclusion Criteria:

* primigravida, singleton pregnancy, maternal age 18-35 years, and pregnancy duration 16-20 weeks at the time of study inclusion.

Exclusion Criteria:

* Women with multi-fetal pregnancy, diabetes mellitus, chronic hypertension, or chronic renal disease

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 1200 (Estimated)
Dates: Start 2016-07-01 (Actual); Primary Completion 2018-08-01 (Estimated); Study Completion 2018-08-01 (Estimated)

PRIMARY OUTCOMES:
Pre eclampsia | after 20 weeks
  develpment of pre eclampsia

SECONDARY OUTCOMES:
preterm labour | less than completed 37 weeks
  early delivery before term

CONTACTS AND LOCATIONS:
Overall Officials: Adel S Salah El-Din, MD, Principal Investigator — Assistant Proffesor
Locations (1):
- Ain Shams University Maternity Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided